CLINICAL TRIAL: NCT04942990
Title: The Effectiveness of Calistenic Exercise Training in Adolescents Receiving Online Education During COVID-19 Pandemic
Brief Title: The Effectiveness of Calistenic Exercise Training in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nihan Ozunlu Pekyavas, Associated Proffesor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KA20/478
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Adolescent Development
Keywords: Adolescent; Teleconference; exercise training; calisthenic exercise; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise training group (Experimental): The duration of the study was targeted as 8 weeks. Our trainings consist of 3 sessions per week, with an average of 45 minutes of calisthenic exercises per session. Exercises initially started with an average of 30 minutes, 10 repetitions, gradually increased difficulty once every two weeks, time increased to 45 minutes movements were modified for those who were forced to perform the exercise program. The program was completed with 5 minutes of warm-up and 5 minutes of cooling exercises before exercise training. All exercises were conducted on a video chat platform supervised by an experienced physiotherapist.
  Interventions: Other: calisthenic exercises
- control group (No Intervention): no exercise was given

INTERVENTIONS:
Other: calisthenic exercises — these exercises are a kind of exercise for increasing cardiovascular endurance
  Arms: exercise training group

SUMMARY:
Objective: The aim of this study is to examine the effectiveness of calisthenic exercise training applied via video chat application on physical activity, physical fitness, quality of life and sleep, and anxiety and depression levels in adolescents during distance education. Material and methods: In our study, 38 adolescents were randomly divided into two equal groups as exercise training group and control group. Calisthenic exercise training was given to the exercise training group for eight weeks, three days a week, via video chat application and under the supervision of a physiotherapist. The control group was evaluated before and after the study period. Physical activity levels of individuals; International Physical Activity Scale, quality of life; Children's Quality of Life Scale, anxiety depression levels; Beck Anxiety Scale, Reynolds Depression Scale and sleep quality were evaluated with Pittsburg Sleep Quality Index.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescent children

Exclusion Criteria:

* Individuals with a disease that could prevent them from doing our exercise training were not included in the study.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
The levels of physical activity | 8 weeks
  International physical Activity Survey: The short form, which has improved Turkish validity and reliability, consists of 7 questions. It provides information about the time spent in severe, moderate walking and sitting activities over the past week. The total calculated energy is calculated as the met spent per minute.
sleep quality | 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) has been used to assess sleep quality. Applied at start-up and end of 8 weeks. PSQI allows him to identify disturbances in the last month of his sleep. It consists of 24 questions in total. Components are a test that evaluates sleep time, delays in sleep, frequency and severity of sleep-related problems and the impact of poor sleep on the individual's life activity
quality of children's lives | 8 weeks
  Pediatric Quality of life Questionniare Short Form (PedsQL-SF) has been used to measure the quality of children's lives. Developed by Varni and his friends in 1999, Memik conducted a study of the validity and reliability of the scale in 2008. the scale of 23 points is scored in three areas. On the scale, scores and total points are calculated in the areas of emotional functionality, social functionality and school functionality. The scale is scored 0,25,50,75,100 points, equal to 4, 3, 2, 1, 0 respectively. Scale total score, physical health total score is calculated individually and bullet points are collected assessing emotional, social, school functionality, resulting in psychosocial health total score. The higher the points total, the better the quality of life is concluded
the level of anxiety | 8 weeks
  The Beck anxiety Scale was used to determine the level of anxiety. It consists of 21 questions in total. Each item is rated between 0-3 and 4. All points are collected and the higher the score, the higher the anxiety severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No